CLINICAL TRIAL: NCT06774768
Title: Use of Machine-learning Algorithms, Biomarkers and Measures of Quality of Life to Personalize Medical Management of Liver and Heart Transplant Recipients
Acronym: DARE
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: DARE; PNC0000002 3000435 (Other Grant/Funding Number: Bando PNRR - Ministero della Salute)
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Artificial Intelligence (AI); Hepatocellular Carcinoma (HCC); Heart Transplantation; Liver Transplantation; Machine Learning; Major Cardiovascular Event
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — All enrolled patients will receive additional blood sampling at enrolment (approximately 20 ml) and then at 6 and 12 month of follow-up, during a venopucture performed for the standard laboratory follow-up. Additional samples will be used for assaying a comprehensive array of biomarkers that may provide information regarding immune system activity (T-regs, circulating nanovescicles, microRNA), graft injury (donor-derived cell free DNA), and susceptibility to infection (Quantiferon Monitor; Torque Teno Virus).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational, low risk tissue based, non-pharmacological, retrospective-prospective study for adults heart and liver transplant patients, related to IRCCS Azienda Ospedaliero-Universitaria di Bologna (IRCCS AOUBO).

This clinical study is part of the national multicentric project DARE. The project has the wide overarching aim to develop digital solutions for personalized healthcare.

DETAILED DESCRIPTION:
This study is structured in two phases: 1) a retrospective phase that aims to develop ML-based scores that can allow to predict at patient level the risk of infections, cardiovascular diseases, new onset malignancies and chronic graft dysfunction, and describing the trajectory of this risk over time; 2) a prospective phase in which we test the association of biomarkers, QoL and frailty assessments with the ML-scores applied prospectively in heart and liver transplant recipients.

ELIGIBILITY:
Retrospective cohort Inclusion criteria Receiving a heart or liver transplantation at IRCCS AOUBO between January 2008 and December 2020.

Surviving at least 6 months after surgery Receiving at least one outpatient clinical assessment, comprising clinical evaluation, standard laboratory tests, and graft ultrasound Older than 18 years old

Exclusion criteria Unavailability of medical records in the standard data repositories of IRCCS AOUBO

Prospective cohort

Inclusion criteria Older thant 18 years old Receiving a heart or liver transplantation at least 6 months before study entry and being in active follow up at IRCCS AOUBO Obtaining informed consent

Exclusion criteria None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the retrospective phase we will include all patients receiving heart or liver transplantation between January 2008 and December 2020 and surviving at least 6 months after surgery.
  In the prospective phase we will consider for enrolment all patients with heart or liver transplantation actively on follow-up at IRCCS AOUBO from January 2024 and January 2026.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-01-30 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Infection | 4 years
  Infection, defined as systemic or organ-specific syndrome characterized by evidence of inflammatory response, abnormal organ function, and need for intravenous antimicrobial treatment, with or without microbiological isolate.
Major Cardiovascular Event (MACE) | 4 years
  Major Cardiovascular Event (MACE) defined as, fatal or non-fatal myocardial infarction, ischemic or hemorrhagic stroke, admission for heart failure, new onset arrhythmia, new onset symptoms for peripheral artery diseases
New onset malignancy | 4 years
  New onset malignancy, defined as hematopoietic or solid malignant neoplasm, developing after transplantation
Chronic graft dysfunction | 4 years
  Chronic graft dysfunction; in HTX recipients defined as onset of one or more of the following: CAV grade 2 or greater as diagnosed by standard of care coronary angiography; diffuse fibrosis with signs of diastolic or systolic left ventricle dysfunction. In LTX we define chronic graft dysfunction as progressive fibrosis, cholestasis and reduced protein synthesis, portal hypertension.

SECONDARY OUTCOMES:
ML-Scores as Surrogate Endpoints | 4 years
  The ML-scores developed to predict the primary outcomes will be used as secondary study outcomes for the prospective phase of the study, and will be tested as surrogate endpoints for clinical outcomes. In this approach, we will analyze the association between such defined surrogate endpoints and biomarkers, QoL and cognitive scores, and frailty measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Luciano Potena, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS - Azienda ospedaliero-universitaria di Bologna, Bologna, Italy